CLINICAL TRIAL: NCT00006249
Title: PEG-Intron Observation After Regional Lymph Node Dissection in AJCC Stage III (TxN1-2MO) Melanoma Patients: a Randomized Phase III Trial
Brief Title: Interferon Alfa Following Surgery in Treating Patients With Stage III Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-18991; EORTC-18991
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Chemotherapy, Adjuvant

ARMS (2):
- observation (No Intervention): 5 years observation + 5 years follow up
- pegylated interferon alfa (Experimental): 5 years pegylated interferon alfa + 5 years follow up
  Interventions: Biological: pegylated interferon alfa; Procedure: adjuvant therapy

INTERVENTIONS:
Biological: pegylated interferon alfa
  Arms: pegylated interferon alfa
Procedure: adjuvant therapy
  Arms: pegylated interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of the cancer cells. It is not yet known if this treatment is more effective than observation following surgery for stage III melanoma.

PURPOSE: Randomized phase III trial to determine the effectiveness of interferon alfa in treating patients who have undergone surgery for stage III melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effect of adjuvant therapy with pegylated interferon alfa vs observation, in terms of distant metastases-free survival, in patients with previously resected stage III melanoma.
* Compare the overall survival in these patients after treatment with pegylated interferon alfa vs observation.
* Determine the toxicity of pegylated interferon alfa in these patients.
* Determine the compliance of these patients treated with pegylated interferon alfa.
* Compare the quality of life in these patients after treatment with pegylated interferon alfa vs observation.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to type of nodal involvement (N1 vs N2), number of positive nodes (1 vs 2-4 vs 5 or more vs not assessed), Breslow primary (T1-2 vs T3 vs T4 vs unknown), ulceration of primary tumor (absent vs present vs unknown), sex, and center. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive pegylated interferon alfa subcutaneously weekly for 5 years.
* Arm II: Patients undergo observation only. Treatment continues in the absence of distant metastases or unacceptable toxicity.

Quality of life is assessed at baseline, and then at months 3, 12, 24, 36, 48, and 60.

Patients are followed every 6 months for 5 years.

PROJECTED ACCRUAL: A total of 1,200 patients (600 per treatment arm) will be accrued for this study within 1.5-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously resected stage III primary cutaneous melanoma or unknown primary with regional lymph node involvement

  * N1 disease

    * Microscopic, nonpalpable nodal involvement
    * Primary melanoma of any stage with clinically inapparent N1 regional lymph node metastases (T1-4, N1, M0) detected by elective lymph node dissection or sentinel node biopsy
  * N2 disease

    * Palpable nodal involvement with synchronous primary melanoma or apparent nodal disease after prior excision (any pT, N2, M0)
  * Regional lymph node recurrence at any interval after surgery for primary melanoma of any depth (T1-4, rN2, M0)
* Complete resection of primary melanoma with adequate surgical margins
* Full lymphadenectomy must be performed within 70 days of study
* No mucous membrane melanoma or ocular melanoma
* No evidence of distant or nonregional lymph node metastases or in transit metastases (even if previously resected)
* No incompletely resected disease due to gross extracapsular extension

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* SGOT and SGPT less than 2 times upper limit of normal
* No active hepatitis

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* No severe cardiovascular disease including the following:

  * Arrhythmias requiring chronic treatment
  * Congestive heart failure (New York Heart Association class III or IV)
  * Symptomatic ischemic heart disease

Other:

* No other prior malignancy within the past 5 years except surgically cured nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No thyroid dysfunction unresponsive to therapy
* No uncontrolled diabetes mellitus
* No active autoimmune disease
* No active and/or uncontrolled infection
* No history of neuropsychiatric disorder requiring hospitalization
* No known active alcohol or drug abuse
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior interferon alfa
* No prior immunotherapy for melanoma
* No other concurrent immunologic or biologic therapy
* No concurrent colony stimulating factors including epoetin alfa and filgrastim (G-CSF)

Chemotherapy:

* No prior chemotherapy for melanoma
* No concurrent chemotherapy

Endocrine therapy:

* No prior hormonal therapy for melanoma
* No concurrent hormonal therapy
* No concurrent chronic systemic corticosteroid therapy

Radiotherapy:

* No prior radiotherapy for melanoma
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* Recovered from any prior recent surgery

Other:

* At least 30 days since other prior experimental therapy
* No other concurrent investigational drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1258 (Actual)
Dates: Start 2000-06; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
distant-metastasis free-survival (DMFS) | from randomization
  distant-metastasis free-survival (DMFS) after randomization

SECONDARY OUTCOMES:
survival | from randomization till death
  duration of survival: time from randomization until death, whatever the cause
toxicity | from randomization
  toxicity

OTHER OUTCOMES:
quality of life | from randomization
  Quality of life evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Alexander M. M. Eggermont, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (104):
- Australia (5):
  - Peter MacCallum Cancer Institute, East Melbourne, Victoria
  - Austin and Repatriation Medical Centre, Heidelberg West, Victoria
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Perth, Western Australia
  - David Maddison Clincial Sciences, Newcastle
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Hopital Universitaire Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Clinique Notre Dame de Grace, Gosselies
  - U.Z. Gasthuisberg, Leuven
- National Centre of Oncology, Sofia, Bulgaria
- University Hospital Sestre Milosrdnice, Zagreb, Croatia
- Charles University Hospital, Prague (Praha), Czechia
- North-Estonian Regional Hospital Cancer Centre, Tallinn, Estonia
- France (23):
  - Centre Hospitalier Universitare d'Amens, Amiens
  - CHR de Besancon - Hopital Saint-Jacques, Besançon
  - Hopital Saint Andre, Bordeaux
  - CHU Ambroise Pare, Boulogne-Billancourt
  - CHR de Grenoble - La Tronche, Grenoble
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Hopital St. Eloi, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Hopital L'Archet - 2, Nice
  - Hopital Bichat - Claude Bernard, Paris
  - Hopital Saint-Louis, Paris
  - Hopital Haut Leveque, Pessac
  - Centre Hospitalier Universitaire, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier Regional et Universitaire de Saint-Etienne, Saint-Priest-en-Jarez
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Centre Hospitalier Regional Metz Thionville, Thionville
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Germany (11):
  - Robert Roessle Klinik, Berlin
  - Saint Josef Hospital, Bochum
  - Stadt. Kliniken, Dortmund
  - Universitaet Erlangen, Erlangen
  - Georg August Universitaet, Göttingen
  - Haematologisch-Onkologische Praxis Altona, Hamburg
  - Universitaets-Hautklinik Heidelberg, Heidelberg
  - Universitaet Leipzig - Chirurgische Klinik und Poliklinik I, Leipzig
  - Otto - Von - Guericke - Universitaet Magdeburg, Magdeburg
  - Klinikum der Stadt Mannheim, Mannheim
  - Universitaet Wuerzburg/Hautkrankheiten, Würzburg
- Israel (3):
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospendale S.M. Annunziata-A.S.DI Firenze, Florence
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - European Institute of Oncology - Chemo Prevention, Milan
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan)
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Istituto Regina Elena, Rome
  - Universita Degli Studi di Torino, Torino
- Netherlands (5):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - Academisch Ziekenhuis Utrecht, Utrecht
- Poland (2):
  - Great Poland Cancer Center, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw
- Portugal (2):
  - Instituto Portugues de Oncologia de Francisco Gentil - Centro de Lisboa, Lisbon
  - Instituto Portugues de Oncologia Centro do Porto, SA, Porto
- Institute of Oncology, Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario, Zaragoza
- Switzerland (4):
  - Kantonspital Aarau, Aarau
  - Inselspital, Bern, Bern
  - Ratisches Kantons und Regionalspital, Chur
  - UniversitaetsSpital, Zurich
- Turkey (Türkiye) (2):
  - Vakif Gureba Training Hospital, Istanbul
  - Ege University Medical School, Izmir
- United Kingdom (26):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Addenbrooke's NHS Trust, Cambridge, England
  - Cheltenham General Hospital, Cheltenham, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Royal Surrey County Hospital, Guildford, England
  - Princess Royal Hospital, Hull, England
  - St. James's Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Saint Bartholomew's Hospital, London, England
  - Royal Free Hospital, London, England
  - Guy's and St. Thomas' Hospitals NHS Trust, London, England
  - St. George's Hospital, London, England
  - Royal Marsden NHS Trust, London, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Salisbury District Hospital, Salisbury, England
  - Weston Park Hospital, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden Hospital, Sutton, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Belfast City Hospital Trust, Belfast, Northern Ireland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Velindre Cancer Center at Velinde Hospital, Cardiff, Wales
  - Selly Oak Hospital at University Hospital NHS Trust, Birmingham
  - Churchill Hospital, Oxford

REFERENCES:
- [Background] Eggermont AM, Suciu S, Testori A, Kruit WH, Marsden J, Punt CJ, Santinami M, Sales F, Schadendorf D, Patel P, Dummer R, Robert C, Keilholz U, Yver A, Spatz A. Ulceration and stage are predictive of interferon efficacy in melanoma: results of the phase III adjuvant trials EORTC 18952 and EORTC 18991. Eur J Cancer. 2012 Jan;48(2):218-25. doi: 10.1016/j.ejca.2011.09.028. Epub 2011 Nov 5. PMID 22056637
- [Result] Eggermont AM, Suciu S, Santinami M, et al.: EORTC 18991 phase III trial: Long-term adjuvant pegylated interferon-α2b (PEG-IFN) versus observation in resected stage III melanoma: long-term results at 7.6-years follow-up. [Abstract] J Clin Oncol 29 (Suppl 15): A-8506b, 2011.
- [Result] Bouwhuis MG, Suciu S, Testori A, Kruit WH, Sales F, Patel P, Punt CJ, Santinami M, Spatz A, Ten Hagen TL, Eggermont AM. Phase III trial comparing adjuvant treatment with pegylated interferon Alfa-2b versus observation: prognostic significance of autoantibodies--EORTC 18991. J Clin Oncol. 2010 May 10;28(14):2460-6. doi: 10.1200/JCO.2009.24.6264. Epub 2010 Apr 12. PMID 20385998
- [Result] Eggermont AM, Bouwhuis MG, Kruit WH, Testori A, ten Hagen T, Yver A, Xu C. Serum concentrations of pegylated interferon alpha-2b in patients with resected stage III melanoma receiving adjuvant pegylated interferon alpha-2b in a randomized phase III trial (EORTC 18991). Cancer Chemother Pharmacol. 2010 Mar;65(4):671-7. doi: 10.1007/s00280-009-1072-z. Epub 2009 Jul 21. PMID 19621225
- [Result] Bottomley A, Coens C, Suciu S, Santinami M, Kruit W, Testori A, Marsden J, Punt C, Sales F, Gore M, Mackie R, Kusic Z, Dummer R, Patel P, Schadendorf D, Spatz A, Keilholz U, Eggermont A. Adjuvant therapy with pegylated interferon alfa-2b versus observation in resected stage III melanoma: a phase III randomized controlled trial of health-related quality of life and symptoms by the European Organisation for Research and Treatment of Cancer Melanoma Group. J Clin Oncol. 2009 Jun 20;27(18):2916-23. doi: 10.1200/JCO.2008.20.2069. Epub 2009 May 11. PMID 19433686
- [Result] Fusi A, Collette S, Busse A, Suciu S, Rietz A, Santinami M, Kruit WH, Testori A, Punt CJ, Dalgleish AG, Spatz A, Eggermont AM, Keilholz U. Circulating melanoma cells and distant metastasis-free survival in stage III melanoma patients with or without adjuvant interferon treatment (EORTC 18991 side study). Eur J Cancer. 2009 Dec;45(18):3189-97. doi: 10.1016/j.ejca.2009.09.004. Epub 2009 Sep 28. PMID 19793643
- [Result] Eggermont AM, Suciu S, Santinami M, Testori A, Kruit WH, Marsden J, Punt CJ, Sales F, Gore M, MacKie R, Kusic Z, Dummer R, Hauschild A, Musat E, Spatz A, Keilholz U; EORTC Melanoma Group. Adjuvant therapy with pegylated interferon alfa-2b versus observation alone in resected stage III melanoma: final results of EORTC 18991, a randomised phase III trial. Lancet. 2008 Jul 12;372(9633):117-126. doi: 10.1016/S0140-6736(08)61033-8. PMID 18620949
- [Result] Eggermont AM, Suciu S, Santinami M, et al.: EORTC 18991: long-term adjuvant pegylated interferon-alpha2b (PEG-IFN) compared to observation in resected stage III melanoma, final results of a randomized phase III trial. [Abstract] J Clin Oncol 25 (Suppl 18): A-8504, 473s, 2007.